CLINICAL TRIAL: NCT04545710
Title: A Phase II Trial of Osimertinib and Abemaciclib With a Focus on Non-Small Cell Lung Cancer Patients With EGFR Activating Mutations With Osimertinib Resistance
Brief Title: Osimertinib and Abemaciclib in EGFR Mutant Non-Small Cell Lung Cancer After Osimertinib Resistance
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Hatim Husain, Associate Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 190752
Record Dates: First submitted 2020-09-04; First posted 2020-09-11 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — abemaciclib; osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single Arm, POC (Experimental): Single arm, POC Safety and Efficacy
  Osimertinib 80 mg QD Abemaciclib 150mg BID
  Interventions: Drug: Abemaciclib; Drug: Osimertinib

INTERVENTIONS:
Drug: Abemaciclib — Abemaciclib 150mg BID
  Other Names: Verzenios
Drug: Osimertinib — Osimertinib 80mg daily
  Other Names: Tagrisso

SUMMARY:
Lung cancer is the leading cause of cancer deaths. Advances in the systemic treatment of non-small cell lung cancer (NSCLC) have increased survival in metastatic EGFR-mutated NSCLC. However resistance to therapy can develop.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer deaths. Advances in the systemic treatment of non-small cell lung cancer (NSCLC) have increased survival in metastatic EGFR-mutated NSCLC. However resistance to therapy can develop.

NSCLC tumors with EGFR-activating mutations are exquisitely sensitive to EGFR tyrosine kinase inhibitors with overall response rates approximating 80%. The third generation EGFR compound osimertinib is a standard first line option. Resistance to the third generation EGFR-TKI osimertinib can develop with a median PFS of 18.9 months. Current research examining acquired resistance to EGFR-TKIs has focused on overcoming these main mechanisms of EGFR-TKI resistance and understanding the impact of co-occurring alterations. Frequently altered pathways concomitantly affected with EGFR in lung cancer are cell cycle genes. This study will explore a strategy to inhibit EGFR and CDK4/6 in resistant EGFR mutated lung cancer patients post progression on osimertinib.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed NSCLC-lung adenocarcinoma histology.
* Tumor must harbor an EGFR activating mutation (Exon 21 L858R, Exon 19 deletion, Exon 18 G719X, Exon 21 L861Q).
* Patient must have Stage IV, recurrent or metastatic disease with EGFR mutant disease.
* Patient must have progressive disease on or after osimertinib (any number of prior treatment is allowed).
* At least one measurable lesion according to RECIST version 1.1
* Age >18 years
* ECOG performance status ≤1
* Patients who received chemotherapy must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] Grade ≤1) from the acute effects of chemotherapy except for residual alopecia or Grade 2 peripheral neuropathy prior to randomization. A washout period of at least 21 days is required between last chemotherapy dose and randomization (provided the patient did not receive radiotherapy).
* Patients who received adjuvant radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of radiotherapy and randomization.

The patient has adequate organ function for all of the following criteria, as defined below.

Table 1: Laboratory Value Guidance to Establish Adequate Organ Function System Laboratory Value Hematologic ANC 1.5 × 109/L Platelets 100 × 109/L Hemoglobin 8 g/dL Patients may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator. Initial treatment must not begin earlier than the day after the erythrocyte transfusion.

Hepatic Total bilirubin 1.5 × ULN Patients with Gilbert's syndrome with a total bilirubin ≤2.0 times ULN and direct bilirubin within normal limits are permitted.

ALT and AST 3 × ULN Renal Serum creatinine 1.5 × ULN

Abbreviations: ALT = alanine aminotransferase; ANC = absolute neutrophil count; AST = aspartate aminotransferase; ULN = upper limit of normal.

* Negative urinary pregnancy test within 7 days prior to entry of study.
* Men and women of child bearing age must agree to contraception methods prior to entry of study and continue on that for 3 months for women and 6 months for men after last dose of osimertinib (details will be submitted in actual protocol) and notification of PI if pregnancy occurs.
* Patients with brain metastases may enroll in this study providing they have been treated and remain asymptomatic.
* The patient is able to swallow oral medications.

Exclusion Criteria:

* Chemotherapy or other investigational agent within three weeks prior to the start of study treatment.
* Radiotherapy within 4 weeks prior to randomization, except as follows:
* Palliative radiation to target organs other than chest or stereotactic radiotherapy to the chest may be allowed up to 2 weeks prior to treatment with osimertinib and abemaciclib.
* Single dose palliative treatment for symptomatic metastasis outside above allowance to be discussed with sponsor prior to enrolling.
* Major surgery within 4 weeks before starting study treatment or scheduled for surgery during the projected course of the study.
* Known hypersensitivity to osimertinib or the excipients of any of the trial drugs.
* History or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure NYHA classification of 3, unstable angina or poorly controlled arrhythmia as determined by the investigator. Myocardial infarction within 6 months prior to study enrollment.
* Women of child-bearing potential (WOCBP) and men who are able to father a child, unwilling to be abstinent or use adequate contraception prior to study entry, for the duration of study participation and for at least 28 days after treatment has ended. <Note: for osimertinib this must be 28 days, however this may be longer for other drugs.
* Female patients of childbearing potential who are nursing or are pregnant or are not using an acceptable method of birth control, or do not plan to continue using this method throughout the study and/or do not agree to submit to pregnancy testing required by this protocol.
* Previous or concomitant malignancies at other sites, except effectively treated non-melanoma skin cancers, carcinoma in situ of the cervix, ductal carcinoma in situ or effectively treated malignancy that has been in remission for more than 3 years and is considered to be cured.
* Known pre-existing interstitial lung disease (patients with previous radiation induced interstitial lung disease are allowed provided they do not require active treatment and symptoms attributed to interstitial lung disease have resolved).
* Any history or presence of poorly controlled gastrointestinal disorders that could affect the absorption of osimertinib (e.g. Crohn's disease, ulcerative colitis, chronic diarrhea, and malabsorption).
* Active hepatitis B infection (defined as presence of HepB sAg and/ or Hep B DNA), active hepatitis C infection (defined as presence of Hep C RNA) and/or known HIV carrier.
* QTcF > 470 ms on average of 3 ECG recordings
* Leptomeningeal carcinomatosis.
* Patients with controlled CNS metastases are allowed. Radiotherapy or surgery for CNS metastases must have been completed >2 weeks prior to study entry. Patients must be neurologically stable, having no new neurologic deficits on clinical examination, and no new findings on CNS imaging. Steroid use for management of CNS metastases must be at a stable dose for two weeks preceding study entry.
* The patient has serious preexisting medical condition(s) that would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
* The patient has active bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive].
* The patient has a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest.
* Clinically active interstitial lung disease, radiation pneumonitis requiring steroid treatment and further entry to be determined on an individual basis.
* Use of medications or supplements known to be major inducers of CYP3A4.
* Comorbidities not limited to unstable angina, congestive heart failure; EKG abnormalities including but not limited to QT prolongation; gastrointestinal diseases limiting absorption of oral medications; psychiatric illnesses and other social situations which may limit participation and compliance on the study.
* Prior CDK4/6 inhibitor treatment is prohibited

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-11-21 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival at 6 months | 6 months
  Rate of Progression Free Survival at 6 months on the combination.

CONTACTS AND LOCATIONS:
Overall Officials: Hatim Husain, MD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Moores Cancer Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No